CLINICAL TRIAL: NCT01520298
Title: Intravenous Acetaminophen as Adjuvant Therapy for Pain Control in Geriatric Hip Fracture Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in recruiting subjects for the trial.
Sponsor: Lancaster General Hospital (Other)
Responsible Party: Principal Investigator, Michael A. Horst, PhD, MPHS, MS, Director of Research, Lancaster General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-52
Record Dates: First submitted 2012-01-23; First posted 2012-01-27 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Pain; Hip Fracture
MeSH Terms: conditions — Pain; Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): For the control group, a total of 100 mLs of 0.9% sodium chloride will be transferred to a Hospira LifeCare container and infused over 15 minutes (6.7 mL/min). A beyond use expiration of 6 hours will be placed on the container.
  Interventions: Drug: Placebo
- Acetaminophen treatment (Active Comparator): For the treatment group, a total of 100 milliliters (mLs) of acetaminophen (1000 mg) will be transferred to a Hospira LifeCare container and infused over 15 minutes (6.7 mLs/min). A beyond use expiration of 6 hours at room temperature will place on the container, as recommended by the manufacturer.
  Interventions: Drug: Acetaminophen IV

INTERVENTIONS:
Drug: Placebo — For the control group, a total of 100 mLs of 0.9% sodium chloride will be transferred to a Hospira LifeCare container and infused over 15 minutes (6.7 mL/min). A beyond use expiration of 6 hours will be placed on the container. All admixture manipulations will be completed by the pharmaceutical staff according to the chapter 797 guidelines in the U.S. Pharmacopoeia. The treatment period will begin after admission and randomization, and will continue until surgical intervention.
  Arms: Placebo
Drug: Acetaminophen IV — For the treatment group, a total of 100 milliliters (mLs) of acetaminophen (1000 mg) will be transferred to a Hospira LifeCare container and infused over 15 minutes (6.7 mLs/min). A beyond use expiration of 6 hours at room temperature will place on the container, as recommended by the manufacturer. All admixture manipulations will be completed by the pharmaceutical staff according to the chapter 797 guidelines in the U.S. Pharmacopoeia. The treatment period will begin after admission and randomization, and will continue until surgical intervention.
  Arms: Acetaminophen treatment

SUMMARY:
This research study is a prospective, randomized, blinded, placebo controlled trial evaluating the benefit of IV acetaminophen (Ofirmev™) as adjuvant analgesia in geriatric hip fracture patients. IV acetaminophen has received FDA approval. IV acetaminophen does not have the liver toxicity as oral acetaminophen. No oral acetaminophen will be administered. All patients diagnosed with a hip fracture aged at least 65 years and expected to undergo surgical intervention are eligible to participate. Hip fractures affect greater than 300,000 geriatric patients annually, representing the second leading cause of hospitalization for this patient population. Pain control in these patients is often problematic due to co-morbidities and changes in their pharmacokinetic and pharmacodynamic profiles. Subjects may receive the normal DVT prophylactic treatments post-op.

DETAILED DESCRIPTION:
Approximately 46 subjects will be enrolled at LGH. Subjects will be randomized 1:1 to receive either IV acetaminophen 1000 mg q6 hours (FDA recommended dose) or IV placebo. While receiving the study drug/placebo the subject's blood pressure, heart rate, respiratory rate, & pain intensity will be monitored. Additional pain meds will be given if needed. Study treatment will continue until subject is taken into the operating room; at that time the intervention will be discontinued and other pain medication will be provided. Participation in the study will end at time of discharge from the hospital. Researchers are expecting a 33% decrease in opioid use for subjects randomized to treatment group.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged at least 65 years with a diagnosis of hip fracture with whom surgical intervention is expected
* Patients with the following surgeons ( David Hughes MD, Gerald Rothacker MD, Frank Essis MD, James Carson MD, Michael Gish MD, Vincent Battista MD)

Exclusion Criteria:

* Documented drug or alcohol addiction or abuse
* Documented serum sodium levels > 145 mmol/L
* Documented serum chloride levels > 107 mmol/L
* Impaired liver function defined as an ALT or AST > 3 times the upper limit of normal, Child-Pugh class C, or patients with documented active liver disease
* Known allergy or intolerance to acetaminophen
* Weight ≤ 50 kg
* Creatinine clearance (CrCl) ≤ 30 ml/min as determined by the Cockcroft-Gault equation
* Documented dementia
* Acetaminophen (> 650 mg) or opioid (> 7 mg IV morphine equivalence) use within the previous 24 hours
* Documented chronic opioid use

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Opioid usage | 24 Hours
  Participants will be assessed for opioid utilization until they go to surgery: an average of 24 hours.

SECONDARY OUTCOMES:
Length of stay | Up to 1 week
  Participants will be followed for the duration of their hospital stay, an expected average of 1 week. Length of stay, vital signs (blood pressure, heart rate, respiratory rate), pain scores using the visual analog scale (VAS), and opioid induced side effects including: nausea, vomiting, changes in blood pressure and delirium
Vital signs | Up to 1 week
  Participants will be followed for the duration of their hospital stay, an expected average of 1 week. Length of stay, vital signs (blood pressure, heart rate, respiratory rate), pain scores using the visual analog scale (VAS), and opioid induced side effects including: nausea, vomiting, changes in blood pressure and delirium
Pain scores | Up to 1 week
  Participants will be followed for the duration of their hospital stay, an expected average of 1 week. Length of stay, vital signs (blood pressure, heart rate, respiratory rate), pain scores using the visual analog scale (VAS), and opioid induced side effects including: nausea, vomiting, changes in blood pressure and delirium
Opioid induced side effects | Up to 1 week
  Participants will be followed for the duration of their hospital stay, an expected average of 1 week. Length of stay, vital signs (blood pressure, heart rate, respiratory rate), pain scores using the visual analog scale (VAS), and opioid induced side effects including: nausea, vomiting, changes in blood pressure and delirium

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Costello, PharmD, Study Chair — Lancaster General Hospital; Gerald W Rothacker, MD, Principal Investigator — Lancaster General Hospital; Jason Hall, PharmD, Principal Investigator — Lancaster General Hospital; Jill Rebuck, PharmD, Principal Investigator — Lancaster General Hospital; Michael A Horst, PhD, Principal Investigator — Lancaster General Hospital; Melody Dillman, RN, Principal Investigator — Lancaster General Hospital; Michael Gish, MD, Principal Investigator — Lancaster General Hospital; Vincent Batista, MD, Principal Investigator — Lancaster General Hospital; James H Carson, MD, Principal Investigator — Lancaster General Hospital; Frank M Essis, MD, Principal Investigator — Lancaster General Hospital; David P Hughes, MD, Principal Investigator — Lancaster General Hospital; Heidi L Testa, RN, Principal Investigator — Lancaster General Hospital; Kay M Knepper, RN, Principal Investigator — Lancaster General Hospital; LouAnne Kruse, RN, Principal Investigator — Lancaster General Hospital
Locations (1):
- Lancaster General Hospital, Lancaster, Pennsylvania, United States

REFERENCES:
- [Background] Abbott C. Falls and hip fractures [updated: February 2011]. University of Missouri-Columbia School of Health Professions. Available at: http://www.vhct.org/case4007/index.htm. Accessed September 26, 2011.
- [Background] Edelstein DM, Aharonoff GB, Karp A, Capla EL, Zuckerman JD, Koval KJ. Effect of postoperative delirium on outcome after hip fracture. Clin Orthop Relat Res. 2004 May;(422):195-200. doi: 10.1097/01.blo.0000128649.59959.0c. PMID 15187857
- [Background] Schuurmans MJ, Duursma SA, Shortridge-Baggett LM, Clevers GJ, Pel-Littel R. Elderly patients with a hip fracture: the risk for delirium. Appl Nurs Res. 2003 May;16(2):75-84. doi: 10.1016/s0897-1897(03)00012-0. PMID 12764718
- [Background] Morrison SR, Magaziner J, McLaughlin MA, Orosz G, Silberzweig SB, Koval KJ, Siu AL. The impact of post-operative pain on outcomes following hip fracture. Pain. 2003 Jun;103(3):303-311. doi: 10.1016/S0304-3959(02)00458-X. PMID 12791436
- [Background] Beaupre LA, Jones CA, Saunders LD, Johnston DW, Buckingham J, Majumdar SR. Best practices for elderly hip fracture patients. A systematic overview of the evidence. J Gen Intern Med. 2005 Nov;20(11):1019-25. doi: 10.1111/j.1525-1497.2005.00219.x. PMID 16307627
- [Background] Baumann T, Strickland J. Pain Management. In:DiPiro JT, et al., editors. Pharmacotherpay. 7th ed. New York: McGraw-Hill;2008. 989-1002
- [Background] Chau DL, Walker V, Pai L, Cho LM. Opiates and elderly: use and side effects. Clin Interv Aging. 2008;3(2):273-8. doi: 10.2147/cia.s1847. PMID 18686750
- [Background] Ofirmev [package insert].San Diego, Ca: Cadence Pharmaceuticals; 2011
- [Background] Sinatra RS, Jahr JS, Reynolds LW, Viscusi ER, Groudine SB, Payen-Champenois C. Efficacy and safety of single and repeated administration of 1 gram intravenous acetaminophen injection (paracetamol) for pain management after major orthopedic surgery. Anesthesiology. 2005 Apr;102(4):822-31. doi: 10.1097/00000542-200504000-00019. PMID 15791113
- [Background] Pettersson PH, Jakobsson J, Owall A. Intravenous acetaminophen reduced the use of opioids compared with oral administration after coronary artery bypass grafting. J Cardiothorac Vasc Anesth. 2005 Jun;19(3):306-9. doi: 10.1053/j.jvca.2005.03.006. PMID 16130055
- [Background] Singla N, Pong A, Newman K; MD-10 Study Group. Combination oxycodone 5 mg/ibuprofen 400 mg for the treatment of pain after abdominal or pelvic surgery in women: a randomized, double-blind, placebo- and active-controlled parallel-group study. Clin Ther. 2005 Jan;27(1):45-57. doi: 10.1016/j.clinthera.2005.01.010. PMID 15763605
- [Background] Cattabriga I, Pacini D, Lamazza G, Talarico F, Di Bartolomeo R, Grillone G, Bacchi-Reggiani L. Intravenous paracetamol as adjunctive treatment for postoperative pain after cardiac surgery: a double blind randomized controlled trial. Eur J Cardiothorac Surg. 2007 Sep;32(3):527-31. doi: 10.1016/j.ejcts.2007.05.017. Epub 2007 Jul 23. PMID 17643995